CLINICAL TRIAL: NCT04577092
Title: Do Motor-cognitive and Motor-motor Dual Task Training Effect Differently Balance Performance in Older Adults?
Brief Title: Dual Task Training for Balance in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aybike Senel, Research Assistant, Sub-investigator, Physiotherapist, MSc, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 13
Record Dates: First submitted 2020-09-25; First posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Geriatrics
MeSH Terms: interventions — Warm-Up Exercise; Cool-Down Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor-Cognitive (Active Comparator): In 10-minute warm up period; neck flexion/extension/side flexion/circumflexion (clockwise and counterclockwise), rounding shoulder back and forth, circumflexion of arm back and forth, side flexion of trunk and rising on the fingertips. After warm up period; participants had been asked to count back from the two-digit number while performing; in standing position, straight walk, side walk, abduction/flexion/extension of hip and hip and knee flexion; in sitting position, hip flexion, knee extension, ankle dorsi - plantar flexion.
  In 10-minute cool down period, stretching of quadriceps femoris muscle, hamstring muscle, achill tendon and cervical muscles were performed.
  Interventions: Other: Warm-up exercise; Other: Motor-Cognitive exercise; Other: Cool-down exercise
- Motor-Motor (Active Comparator): In 10-minute warm up period; neck flexion/extension/side flexion/circumflexion (clockwise and counterclockwise), rounding shoulder back and forth, circumflexion of arm back and forth, side flexion of trunk and rising on the fingertips. After warm up period; participants had been asked to hold with both hand half-filled glasses with 90 degree of flexion elbow and near the trunk while performing; in standing position, straight walk, side walk, abduction/flexion/extension of hip and hip and knee flexion; in sitting position, hip flexion, knee extension, ankle dorsi - plantar flexion. In cool down period, stretching of quadriceps femoris muscle, hamstring muscle, achill tendon and cervical muscles were performed.
  Interventions: Other: Warm-up exercise; Other: Motor-Motor exercise; Other: Cool-down exercise

INTERVENTIONS:
Other: Warm-up exercise — In 10-minute warm up period; neck flexion/extension/side flexion/circumflexion (clockwise and counterclockwise), rounding shoulder back and forth, circumflexion of arm back and forth, side flexion of trunk and rising on the fingertips.
Other: Motor-Cognitive exercise — After warm up period; participants had been asked to count back from the two-digit number while performing; in standing position, straight walk, side walk, abduction/flexion/extension of hip and hip and knee flexion; in sitting position, hip flexion, knee extension, ankle dorsi - plantar flexion.
  Arms: Motor-Cognitive
Other: Motor-Motor exercise — participants had been asked to hold with both hand half-filled glasses with 90 degree of flexion elbow and near the trunk while performing; in standing position, straight walk, side walk, abduction/flexion/extension of hip and hip and knee flexion; in sitting position, hip flexion, knee extension, ankle dorsi - plantar flexion.
  Arms: Motor-Motor
Other: Cool-down exercise — In 10-minute cool down period, stretching of quadriceps femoris muscle, hamstring muscle, achill tendon and cervical muscles were performed.

SUMMARY:
Dual task training (DTT) have been showed that have satisfying effects on older adults. The aim of this study was to compare the effect of motor-cognitive DTT (mCdtt) and motor-motor DTT (mMdtt) on balance, fear of falling, walking functionality and muscle strength in older adults. The participants were divided into two groups; who received mCdtt (Group 1) and who received mMdtt (Group 2). The intervention program had lasted for 8 weeks.

DETAILED DESCRIPTION:
Dual task training (DTT) have been showed that have satisfying effects on older adults. The aim of this study is comparing the effect of motor-cognitive DTT (mCdtt) and motor-motor DTT (mMdtt) on balance, fear of falling, walking functionality and muscle strength in older adults. A total of 50 participants aged 60 and over (mean age: 67.72±7.33 years), having a score ≥ 24 on the Mini-Mental State Exam (MMSE), being in category of walking ability ≥ 4 according to the Functional Ambulation Category (FAC), having no problem in visual ability and hearing were included for this study. The participants who received mCdtt (Group 1) counted back from the two-digit number and the participants who received mMdtt (Group 2) held half-filled glasses with 90o flexion elbow with both hand while performing exercises. The intervention program had lasted for 8 weeks. To assess balance, fear of falling, walking functionality and muscle strength of participants, Berg Balance Scale (BBS), Falls Efficacy Scale International (FES-I), Timed Up and Go (TUG) and Hand-held dynamometer were used, respectively.

ELIGIBILITY:
Inclusion Criteria:

* (1) age over 60 years old
* (2) score ≥ 24 on the Mini-Mental State Exam
* (3) category of walking ability ≥ 4 according to the Functional Ambulation Category
* (4) no problem in visual ability and hearing

Exclusion Criteria:

* (1) a history of specific balance problems (i.e., diagnosed neurological, musculoskeletal or vestibular disorder)
* (2) history of cerebrovascular occasion
* (3) history of hip-knee surgery
* (4) use of medication(s) such as sedatives and hypnotics, antidepressants and benzodiazepines.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-03-18 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | baseline (first assessment)
  BBS is a widely used, reliable and valid scale, which was developed to measure balance in older adults with functional postures and movements. It consists of 14 items scoring from 0 (unable/unsafe) to 4 (independent/safe). The highest score was 56 and means the best ability of balance. Score of 0-20, 21-40 and 41-56 mean bad, fair and good ability of balance, respectively
Berg Balance Scale (BBS) | End of the training (8 weeks after)
  BBS is a widely used, reliable and valid scale, which was developed to measure balance in older adults with functional postures and movements. It consists of 14 items scoring from 0 (unable/unsafe) to 4 (independent/safe). The highest score was 56 and means the best ability of balance. Score of 0-20, 21-40 and 41-56 mean bad, fair and good ability of balance, respectively

SECONDARY OUTCOMES:
Falls Efficacy Scale International (FES-I) | baseline (first assessment)
  FES-I evaluates concerns about falling with 16 items consisting of social and physical activities. Each item can be replied as 1=not all concerned, 2=somewhat concerned 3=fairly concerned and 4=very concerned. Total score is in a range between 16 and 64, a higher score means higher concern about falling.
Falls Efficacy Scale International (FES-I) | End of the training (8 weeks after)
  FES-I evaluates concerns about falling with 16 items consisting of social and physical activities. Each item can be replied as 1=not all concerned, 2=somewhat concerned 3=fairly concerned and 4=very concerned. Total score is in a range between 16 and 64, a higher score means higher concern about falling.
Timed Up and Go (TUG) | baseline (first assessment)
  (TUG) test is a common, simple and quick test for the function, balance, gait and risk of fall assessment. The TUG was showed to be the most evidence-supported functional measure to evaluate risk of falls in older adults. To perform the test, the participants were asked to seat armchair with back support which was 46 cm above from the floor. The participants were instructed to stand up, walk a distance of 3 meters away from the seat as fast as possible, turn, walk back to seat and sit down. The time passed during this maneuver was recorded as seconds with a chronometer.
Timed Up and Go (TUG) | End of the training (8 weeks after)
  (TUG) test is a common, simple and quick test for the function, balance, gait and risk of fall assessment. The TUG was showed to be the most evidence-supported functional measure to evaluate risk of falls in older adults. To perform the test, the participants were asked to seat armchair with back support which was 46 cm above from the floor. The participants were instructed to stand up, walk a distance of 3 meters away from the seat as fast as possible, turn, walk back to seat and sit down. The time passed during this maneuver was recorded as seconds with a chronometer.
Muscle Testing (MT) | baseline (first assessment)
  MT was performed with Hand-held dynamometer (Lafeyette Instrument®, Lafeyette, IN) to assess power and ability for stability, in this study. Antigravity muscles (m. gluteus maximus, m. quadriceps femoris, m. gastrocnemius and m. tibialis anterior) were assessed while performing maximal volunteer isometric contraction (MVIC) and values were recorded as kg. N-1.
Muscle Testing (MT) | End of the training (8 weeks after)
  MT was performed with Hand-held dynamometer (Lafeyette Instrument®, Lafeyette, IN) to assess power and ability for stability, in this study. Antigravity muscles (m. gluteus maximus, m. quadriceps femoris, m. gastrocnemius and m. tibialis anterior) were assessed while performing maximal volunteer isometric contraction (MVIC) and values were recorded as kg. N-1.

OTHER OUTCOMES:
Charlson Comorbidity Index (CCI) | baseline (first assessment)
  CCI was used to measure the comorbidity status of participants. It investigates existence of 17 comorbidities. The final score indicates disease burden and is a good estimator of mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Hanifegul Taskiran, PT, Prof, Study Director — Istanbul Aydın University
Locations (1):
- Istanbul Aydin University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akin H, Senel A, Taskiran H, Kaya Mutlu E. Do motor-cognitive and motor-motor dual task training effect differently balance performance in older adults? Eur Geriatr Med. 2021 Apr;12(2):371-378. doi: 10.1007/s41999-020-00434-8. Epub 2021 Jan 3. PMID 33389715